CLINICAL TRIAL: NCT05819125
Title: Comparison of the Risk of Venous Thromboembolism and Bleeding Events in a Population of Obese Patients Receiving Higher-Dose or Extended-Duration Versus Conventional-Dose or Conventional-Duration of Prophylaxis With Enoxaparin
Brief Title: Comparison of the Risk of Venous Thromboembolism (i.e., Blood Clots in the Veins) and Bleeding Events in a Population of Obese Patients Receiving Higher-Dose or Extended-Duration Versus Conventional-Dose or Conventional-Duration of Prophylaxis (i.e., Preventive Treatment) With Enoxaparin
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision. Termination decision unrelated to safety profile.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: CEF0112; U1111-1288-8394 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Conventional prophylaxis: Hospitalized obese participants with an acute medical condition or undergoing surgery, receiving conventional (i.e., 40 mg once daily for 7 days) enoxaparin VTE prophylaxis
- High dose prophylaxis: Hospitalized obese participants with an acute medical condition or undergoing surgery, receiving high dose enoxaparin for the conventional VTE prophylaxis duration
- Extended duration prophylaxis: Hospitalized obese participants with an acute medical condition or undergoing surgery, receiving the conventional enoxaparin dose for an extended VTE prophylaxis duration
- High dose and extended duration prophylaxis: Hospitalized obese participants with an acute medical condition or undergoing surgery, receiving high dose enoxaparin for an extended VTE prophylaxis duration

SUMMARY:
In individuals with obesity, the optimal dosing and duration of venous thromboembolism (VTE) prophylaxis in settings representing acute medical illness or surgery is limited due to lack of randomized controlled trials (RCTs) focusing specifically on this population. Evidence suggests that in obese participants, both higher dosing and duration of VTE prophylaxis with Low Molecular Weight Heparins (LMWH) may be required to achieve a therapeutic effect similar to non-obese participants.

This non-interventional study utilizes data already collected from a usual clinical practice setting in the Optum US clinical database, representing obese participants hospitalized with an acute medical condition or undergoing surgery receiving enoxaparin prophylaxis. Its aim is to compare the impact of the following enoxaparin prophylaxis strategies on the incidence of symptomatic VTE and major bleeding in the overall study population and prespecified subgroups:

* High versus conventional dose
* Extended versus conventional duration
* Combined High-Dose and Extended-Duration versus Conventional-Dose and Conventional-Duration.

The first date of enoxaparin prophylaxis will be the index date.

DETAILED DESCRIPTION:
The study period will be from February 2010 to September 2021. Participants will be followed for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Medical Patients: Hospitalization due to:

  * Heart failure
  * Ischemic stroke
  * Respiratory insufficiency
  * Infection
  * Inflammatory diseases
  * Active cancer
* Surgical Patents: Following surgery types:

  * Orthopedic
  * Thoracic
  * Abdominal/Pelvic
* Other inclusion criteria:

  * Initiation of enoxaparin prophylaxis (index date)
  * Age ≥ 40 years
  * Body Mass Index (BMI) ≥ 30

Exclusion Criteria:

* VTE or bleeding event during or 3 months prior to index date
* Surgery within 3 months prior to and up to two days following index date
* Atrial fibrillation
* Antiplatelet or anticoagulation therapy within [-32, -2] days before index date
* Chronic Kidney Disease (CKD) stages IV and V, or dialysis
* Pregnancy

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized obese participants with an acute medical condition or undergoing surgery receiving enoxaparin prophylaxis in the Optum Market Clarity database representing integrated information from electronic health records (EHRs) and claims.
Sampling Method: Non-Probability Sample
Enrollment: 21000 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of symptomatic VTE, from index date to Day 90 | Retrospective data analysis from February, 2010 to September, 2021, with this endpoint evaluated up to 90 days after the individual participant's index date.
  The VTE endpoint is intended to represent a new onset symptomatic VTE event. It will be identified in the proposed database by utilizing an algorithm based on the International Classification of Disease 10th and 9th revisions (ICD-10 and ICD-9) codes.
Change in the incidence of major bleeding, from index date to Day 90 | Retrospective data analysis from February, 2010 to September, 2021, with this endpoint evaluated up to 90 days after the individual participant's index date.
  The major bleeding event will be identified via an algorithm based on the International Classification of Disease-10th revision and 9th revision (ICD-10 and ICD-9) codes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi U.S., Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org